CLINICAL TRIAL: NCT00891605
Title: A Phase 1 Safety and Pharmacokinetic Study of ABT-263 in Combination With Paclitaxel in the Treatment of Subjects With Solid Tumors
Brief Title: Safety Study of ABT-263 in Combination With Paclitaxel in Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M10-589
Record Dates: First submitted 2009-04-29; First posted 2009-05-01 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2012-06

CONDITIONS: Solid Tumors
Keywords: Paclitaxel; Solid Tumors
MeSH Terms: interventions — navitoclax; Paclitaxel

ARMS (1):
- Paclitaxel and ABT-263 (Experimental)
  Interventions: Drug: ABT-263; Drug: paclitaxel

INTERVENTIONS:
Drug: ABT-263 — 150 mg of ABT-263 is taken orally once daily on Days 1-3 out of each 21 day cycle. This is a dose escalation study, therefore the dose of ABT-263 will change throughout the study.
  Other Names: Navitoclax
Drug: paclitaxel — 175 mg/m2 over 3 hours of paclitaxel will be given by intravenous infusion on Day 1 of each 21 day cycle.
  Note - The dose and schedule is subject to change based on the toxicities observed.
  Other Names: Taxol

SUMMARY:
Safety study of ABT-263 in Combination with Paclitaxel in Subjects with Solid Tumors.

DETAILED DESCRIPTION:
A Phase 1 Safety and Pharmacokinetic Study of ABT-263 in Combination with Paclitaxel in the Treatment of Subjects with Solid Tumors.

ELIGIBILITY:
Inclusion Criteria

1. Subject must be greater than or equal to 18 years of age.
2. Subject must have a histologically and/or cytologically documented cancer for which paclitaxel has been determined an appropriate therapy, per the Investigator.
3. Subjects with brain metastases must have clinically controlled neurologic symptoms, defined as surgical excision and/or radiation therapy followed by 21 days of stable neurologic function and no evidence of CNS disease progression as determined by CT or MRI within 28 days prior to the first dose of study drug.
4. Subject has an Eastern Cooperative Oncology Group (ECOG) score of less than or equal to 1.
5. Subject must have adequate bone marrow, renal and hepatic function per protocol defined local laboratory testing parameters.

Exclusion Criteria

1. The subject has an underlying, predisposing condition of bleeding or currently exhibits signs of bleeding. The subject has a recent history of thrombocytopenia associated with bleeding within 1 year prior to first dose of study drug.
2. Subject is currently receiving or requires anticoagulation therapy (e.g., warfarin at any dose) or any drugs or herbal supplements that affect platelet function, with the exception of low-dose anticoagulation medications such as heparin that are used to maintain the patency of a central intravenous catheter.
3. The subject has active peptic ulcer disease or other potentially hemorrhagic esophagitis/gastritis.
4. The subject has active immune thrombocytopenic purpura (ITP), autoimmune hemolytic anemia (AIHA), or a history of being refractory to platelet transfusions (within 1 year prior to the first dose of study drug).
5. The subject has a significant history of cardiovascular (e.g., MI, thrombotic or thromboembolic event in the last 6 months), renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, or hepatic disease that in the opinion of the investigator would adversely affect his/her participating in this study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Safety Assessment | Weekly
  Evaluate safety at the defined recommended Phase 2 dose (RPTD) and schedule of ABT-263 in combination with Paclitaxel
Efficacy Assessment | Bi-monthly
  Evaluate preliminary data regarding objective response rate (ORR), progression free survival (PFS), time to tumor progression (TTP), overall survival (OS), duration of overall response, and, ECOG performance status

CONTACTS AND LOCATIONS:
Overall Officials: Mack Mabry, MD, Study Director — Abbott

REFERENCES:
- [Result] Vlahovic G, Karantza V, Wang D, Cosgrove D, Rudersdorf N, Yang J, Xiong H, Busman T, Mabry M. A phase I safety and pharmacokinetic study of ABT-263 in combination with carboplatin/paclitaxel in the treatment of patients with solid tumors. Invest New Drugs. 2014 Oct;32(5):976-84. doi: 10.1007/s10637-014-0116-3. Epub 2014 Jun 5. PMID 24894650